CLINICAL TRIAL: NCT02555475
Title: The Prime Study - Comparing Hepatitis C Care and Treatment in a Primary Health Care Service With a Tertiary Hospital: a Randomised Trial
Brief Title: The Prime Study - Comparing Hepatitis C Care and Treatment in a Primary Health Care Service With a Tertiary Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Macfarlane Burnet Institute for Medical Research and Public Health Ltd (Other)
Collaborators: St Vincent's Hospital Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HREC/15/SVHM/41
Record Dates: First submitted 2015-09-17; First posted 2015-09-21 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2017-07

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; primary care
MeSH Terms: conditions — Hepatitis C | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1, tertiary hospital based care (No Intervention): Group 1: (n=190) Following their initial screen, these participants will be referred to a tertiary hospital for hepatitis C care, transient elastography and DAA treatment (traditional / standard model of care).
- Group 2, community based care (Experimental): Group 2: (n=190) Following their initial screen, these participants will be offered community based hepatitis C care and treatment. Hepatitis C care, transient elastography and DAA treatment will be delivered at the primary healthcare centre only.
  Interventions: Other: community based hepatitis C care and treatment

INTERVENTIONS:
Other: community based hepatitis C care and treatment
  Arms: Group 2, community based care

SUMMARY:
The Prime Study is a randomised trial investigating models of care for hepatitis C in the era of direct acting antiviral (DAA) therapy. The study aims to compare outcomes of hepatitis C care and DAA treatment provided in a primary health care service with a tertiary hospital.

DETAILED DESCRIPTION:
This open label randomised trial will investigate the efficacy of treating people with G1 HCV with DAA in primary healthcare services compared with tertiary hospital clinics. Three hundred and eighty G1 HCV infected patients attending study primary healthcare centres will be invited to participate in the study.

At the primary healthcare centre participants will be randomly allocated to two groups:

Group 1: (n=190) Following their initial screen, these participants will be referred to a tertiary hospital for transient elastography and DAA treatment (traditional model of care)

Group 2: (n=190) Following their initial screen, these participants will be offered transient elastography and DAA treatment delivered at the primary healthcare service only.

Treatment will consist of fixed dose combination paritaprevir, ombitasvir and ritonavir packaged together with dasabuvir, known as Viekira Pak, +/- weight based ribavirin. As cirrhotic patients will be excluded from the study, the duration of treatment is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years;
* Attendance at a study PHCS defined as; Attended appointment at PHCS at least once in 2014 or; Attended at least one consultation with a study community hepatitis nurse between 2012-2014
* Evidence of chronic G1 HCV infection (HCV antibody positive for > 6 months and HCV RNA positive);
* Absence of cirrhosis defined as one of the following:

Liver biopsy within 24 months prior to screening demonstrating absence of cirrhosis (e.g. a Metavir score of 3 or less or an Ishak score of 4 or less); or A screening FibroScan result of <9.6 kPa; or if a FibroScan is unsuccessful A screening Aspartate Aminotransferase to Platelet Ratio Index (APRI) ≤ 2 and no clinical or laboratory evidence of cirrhosis;

* HCV treatment naive or pegylated or standard interferon and ribavirin experienced;
* Willing and able to provide written informed consent

Subjects must have the following laboratory parameters at screening:

* ALT ≤ 10 times the upper limit of normal (ULN);
* AST ≤ 10 times ULN
* Haemoglobin ≥ 12g/dL for males; ≥ 11g/dL for female subjects;
* Platelet count ≥ laboratory lower limit of normal;
* INR ≤ laboratory upper limit of normal, unless stable on an anticoagulant regimen affecting INR;
* Albumin ≥ laboratory lower limit of normal;
* Direct bilirubin ≤ laboratory upper limit of normal;
* Creatinine clearance (Clcr) ≥ 60mL/min as calculated by Cockcroft-Gault equation.

Exclusion Criteria:

* Known cirrhosis defined as:

Liver biopsy within 24 months prior to screening demonstrating cirrhosis (e.g. a Metavir score > 3 or an Ishak score > 4); or A FibroScan result of >12.5 kPa; or Prior clinical evidence of cirrhosis or portal hypertension (i.e. ascites, varices).

* Prior exposure to HCV DAA protease inhibitors
* Currently receiving HCV treatment;
* Testing positive for HIV;
* Testing positive for HBsAg;
* HCC;
* Pregnancy or breastfeeding at screening or baseline;
* Evidence of any condition, therapy, laboratory abnormality or other circumstance (current or prior) that may confound the study's results, or interfere with participation for the full duration of the study, such that it is not in the best interest of the participant;
* Use of concomitant medications that are contraindicated with Viekira Pak within 28 days of the baseline/day 1 visit, that are unable to be ceased for the duration of treatment.

Additional exclusion criteria for participants receiving ribavirin:

* increased baseline risk for anaemia (i.e. history of thalassaemia, spherocytosis, history of GI bleeding) or;
* patients for whom anaemia would be medically problematic or;
* documented of presumed coronary artery disease or cerebrovascular disease, if in the judgement of the investigator, an acute decrease in haemoglobin by up to 4 g/dL (as may be seen with ribavirin) would not be well tolerated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
To measure the proportion of people attending at a Primary Health Care Service for their genotype 1 HCV infection who commence antiviral treatment (Viekira Pak and ribavirin) and have a SVR 12. | Sustained virology response (SVR) rates at week 12 post treatment.

SECONDARY OUTCOMES:
To measure the proportion of people attending a PHCS with G1 HCV infection who commence antiviral treatment (Viekira Pak and ribavirin) if they are managed at a PHCS compared to those who are referred to and managed at a tertiary hospital. | Treatment uptake within 8 weeks of randomisation
To measure the proportion of people with G1 HCV who have an SVR12 at a PHCS compared a tertiary hospital. | SVR rate at week 12 post treatment
To measure the reduction in HCV viraemia (community viral load) among participants considering retention through the cascade of care and SVR12. | up to 24 weeks post treatment
To measure the cost effectiveness of managing and treating people in a primary health service compared to a tertiary hospital. | up to 24 weeks post treatment
To define the cascade of care for patients referred to a community hepatitis nurse for assessment of HCV. | up to 12 weeks post treatment

CONTACTS AND LOCATIONS:
Locations (8):
- Australia (2):
  - St Vincents Hospital Melbourne, Melbourne, Victoria
  - Burnet Institute, Melbourne, Victoria
- New Zealand (6):
  - Hospital Liver Clinic, Greenlane, Auckland
  - Auckland Opioid Treatment Service (AOTS), Point Chevalier, Auckland
  - Hepatitis C Community Clinic, Sydenham, Christchurch
  - Calder Centre Auckland, Auckland
  - Auckland Central liver Clinic, Auckland
  - Community Alcohol and Drug Services, Auckland

REFERENCES:
- [Derived] Wade AJ, Doyle JS, Gane E, Stedman C, Draper B, Iser D, Roberts SK, Kemp W, Petrie D, Scott N, Higgs P, Agius PA, Roney J, Stothers L, Thompson AJ, Hellard ME. Outcomes of Treatment for Hepatitis C in Primary Care, Compared to Hospital-based Care: A Randomized, Controlled Trial in People Who Inject Drugs. Clin Infect Dis. 2020 Apr 15;70(9):1900-1906. doi: 10.1093/cid/ciz546. PMID 31233117
- [Derived] Wade AJ, Doyle JS, Gane E, Stedman C, Draper B, Iser D, Roberts SK, Kemp W, Petrie D, Scott N, Higgs P, Agius PA, Roney J, Stothers L, Thompson AJ, Hellard ME. Community-based provision of direct-acting antiviral therapy for hepatitis C: study protocol and challenges of a randomized controlled trial. Trials. 2018 Jul 16;19(1):383. doi: 10.1186/s13063-018-2768-3. PMID 30012192